CLINICAL TRIAL: NCT07213063
Title: Effects of Chronic Creatine and Beta-Hydroxy-Beta-Methylbutyrate Supplementation on Oxidative Stress, Inflammation, Muscle Strength, and Body Composition in Individuals With Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Collaborators: European University Miguel de Cervantes (Other)
Responsible Party: Principal Investigator, MARIA MARTINEZ, Principal Investigator, Universidad de Burgos
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CreatineSDown.
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Down Syndrome (DS); Supplementation
Keywords: creatine; down syndrome; bone mineral health
MeSH Terms: conditions — Down Syndrome | interventions — Nutrition Assessment; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Active Comparator): Participants will receive placebo supplementation
  Interventions: Other: Nutrition education; Dietary Supplement: Placebo
- Supplementation (Experimental): Participants will receive creatine monohydrate and beta-hydroxy-beta-methylbutyrate supplementation
  Interventions: Other: Nutrition education; Dietary Supplement: Supplement

INTERVENTIONS:
Other: Nutrition education — Participants and their families will also take part in nutrition education sessions to promote healthy eating and lifestyle habits.
Dietary Supplement: Supplement — Supplementation with 3 g/day of creatine monohydrate abd 3 g/day of beta-hydroxy-beta-methylbutyrate for 8 weeks
  Arms: Supplementation
Dietary Supplement: Placebo — Supplementation with 6 g/day of inulin orally for 8 weeks
  Arms: Placebo

SUMMARY:
Purpose:

This study will test whether 8 weeks of creatine and HMB supplementation can improve muscle strength, body composition, balance, and overall health in people with Down syndrome. Participants will also receive nutrition tips during the study.

Who can participate:

People with Down syndrome who can perform basic physical tasks. Must provide consent from the participant and legal guardian.

What participants will do:

Take creatine (3 g/day) and HMB (3 g/day) or placebo for 8 weeks. Complete tests for muscle strength, balance, and cognitive function. Undergo body composition scans and give blood samples for health markers.

Timing:

All tests and blood samples are taken before and after each 8-week period.

Importance:

Results will help determine if creatine and HMB can safely improve strength, balance, and overall health in people with Down syndrome.

DETAILED DESCRIPTION:
This study is an 8-week randomized, placebo-controlled, crossover trial designed to evaluate the effects of daily supplementation with creatine monohydrate (3 g) and beta-hydroxy-beta-methylbutyrate (HMB, 3 g) on body composition, muscle strength, balance, cognitive function, and biomarkers of oxidative stress and inflammation in individuals with Down syndrome. Participants will receive nutritional education throughout the intervention to support a balanced diet.

Primary outcomes include lean mass measured by dual-energy X-ray absorptiometry (DXA).

Secondary outcomes include fat-free mass (bioimpedance), bone mineral density (DXA), handgrip strength, lower limb strength (Five Times Sit-to-Stand Test), upper and lower body isometric strength (K-Pull test), balance (4-Stage Balance Test), and cognitive function assessed by the Timed Up and Go Dual Task. Blood biomarkers of oxidative stress and inflammation, including reduced glutathione (GSH), superoxide dismutase (SOD), C-reactive protein (CRP), interleukins (IL-1, IL-6, IL-7), and tumor necrosis factor-alpha (TNF-α), will be assessed before and after each supplementation period.

All assessments will be performed at baseline and at the end of each 8-week supplementation phase, allowing for evaluation of both physiological and functional responses to creatine and HMB supplementation in this population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Medical confirmation of Down syndrome (trisomy of chromosome 21).
* Physical capacity: Ability to perform basic physical tests (e.g., standing up from a chair or walking without assistance).
* Informed consent: Informed consent will be obtained from both the participant and their legal representative, in compliance with current legislation for individuals requiring support measures.

Exclusion Criteria:

* Chronic kidney disease: Diagnosis of chronic kidney disease.
* Severe motor limitations: Inability to perform the required physical tests (e.g., paralysis or mobility impairments preventing the execution of muscle strength assessments).
* Participation in other studies: Participation in another nutritional or supplementation intervention study within the last 6 months.
* Allergies or intolerances: Known allergy to creatine or to components of the placebo (inulin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Lean mass | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Lean mass (kg) will be evaluated using dual-energy X-ray absorptiometry (DXA): GE Lunar Prodigy DXA device (GE Healthcare, Madison, WI, USA; Encore software version).

SECONDARY OUTCOMES:
Handgrip strength | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Handgrip strength (kg) will be assessed using a handgrip dynamometer.
Bone mineral density | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Total bone mineral density (g/cm2) will be evaluated using dual-energy X-ray absorptiometry (DXA): GE Lunar Prodigy DXA device (GE Healthcare, Madison, WI, USA; Encore software version).
Reduced glutathione (GSH). | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Blood samples will be collected to assess levels of reduced glutathione (GSH).
C-reactive protein (CRP) | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Blood samples will be collected to assess levels of inflammation including C-reactive protein (CRP).
Superoxide dismutase (SOD) activity. | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Blood samples will be collected to assess levels of superoxide dismutase (SOD) activity.
Blood levels of interleukins (IL-1, IL-6, IL-7). | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Blood samples will be collected to assess levels of interleukins (IL-1, IL-6, IL-7).
Tumor necrosis factor-alpha (TNF-α). | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Blood samples will be collected to assess levels of tumor necrosis factor-alpha (TNF-α).
Fat-free mass | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Fat free mass (kg) will be analysed using bioimpedance: InBody S10.
Lower limb strength | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Lower limb strength will be assessed using the Five Times Sit-to-Stand Test (5xSTS), which involved recording the time taken to rise from a 45 cm highchair five times as quickly as possible without using the arms for support.
Balance | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Balance will be using the 4-Stage Balance Test. It involves holding four progressively difficult positions for at least 10 seconds each:
  Feet together: 1 point if the position is held for 10 seconds or more. Partial semi-tandem: 1 point if the position is held for 10 seconds or more.
  Semi-tandem:
  * 2 points: If the position is held for more than 10 seconds.
  * 1 point: If the position is held for between 3 and 9.99 seconds.
  * 0 points: If the position is held for less than 3 seconds. The score ranges from 0 to 4 (best balance).
Cognitive function | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  Cognitive function will be assessed with Timed Up and Go Dual Task (TUGdt) test.
  The participant first performs the Timed Up and Go (TUG) test alone, standing up from a chair, walking a short distance (3 meters) turning, and sitting back down, while simultaneously naming animals within a 10-second period, which assesses verbal fluency.
  The time taken to complete these distances will be recorded, and the fluency in naming the animals will be assessed.
Isometric lower body strength | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  The K-Pull test will be used to evaluate isometric lower body strength
  Participants will perform a seated knee extension test, pushing their leg against the dynamometer with maximal effort. Participants will exert their maximum force against the unyielding device for 3-5 seconds. The peak force achieved (in Newtons) over a minimum of two trials will be recorded
Isometric upper body strength | Baseline (within 2 days before starting supplementation) and at 8 weeks (end of supplementation)
  The K-Pull test will be used to evaluate isometric upper body strength
  Participants will stand with their back against a wall to stabilize the torso. The participant will be instructed to exert a maximal force by pushing their arm outward against the device for 3-5 seconds.The peak force achieved (in Newtons or kilograms-force) over a minimum of two trials will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Burgos, Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No